CLINICAL TRIAL: NCT04271774
Title: Genome Environment Microbiome and Metabolome in Autism
Brief Title: Genome Environment Microbiome and Metabolome in Autism Study
Acronym: GEMMA
Status: Active, not recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Azienda Sanitaria Locale Salerno (Other); National University of Ireland, Galway, Ireland (Other)
Responsible Party: Principal Investigator, Alessio Fasano, Division Chief of Pediatric Gastroenterology and Nutrition, Massachusetts General Hospital
Other Study IDs: 2018P002109
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Autism Spectrum Disorder
Keywords: autism; microbiome; infants; pregnancy; genetic
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Periodic collection of blood, stool, urine and saliva samples from enrolled infant.
  One-time collection of blood, stool, urine and saliva samples from enrolled infant's ASD sibling and parent(s).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants with ASD-affected sibling: Infants, enrolled at 0-6 months of age, who have a sibling diagnosed with ASD.

SUMMARY:
GEMMA is a multicenter longitudinal observational study that follows children who are genetically at-risk of developing autism for their first three years of life, seeking to identify potential biomarkers predictive of autism development in the blood, stool, urine and saliva. The biomarkers identified in this project will contribute to a better understanding of the pathogenesis of ASD in at-risk children and possible solutions for alleviating and/or preventing ASD and ASD-related symptoms in patients in the future.

DETAILED DESCRIPTION:
The GEMMA study will address genomic, environmental, microbiome, and metabolomic factors that may affect the development of autism spectrum disorders (ASD).

Genome: The project will study children who have a first-degree relative (sibling) with ASD so that investigators can understand how their genes may contribute to whether they develop ASD or not. A number of genetic variants identified to date occur in genes encoding glycosylated extracellular proteins and in enzymes directly involved in glycosylation. Investigators will perform whole genome sequencing in the subgroup of children that will develop ASD in order to learn more about these specific genes and also to identify other genes that may be involved in ASD pathogenesis. The genetic variant landscape will be mapped and variants will be annotated and interpreted based on all contextual information available. This effort will enable the identification of patient- and cohort-specific variations that can then be further refined into biomarker signatures and optimized into predictive and diagnostic markers of ASD.

Environment: When infants enroll in the study, investigators will record information about their environment including whether they were born vaginally or by Cesarean section and whether they have received antibiotics. Over time, investigators will also consider other parts of the infant's medical, dietary and social history including feeding modality (breastfeeding versus formula feeding), illnesses, infections, antibiotic use, diet and growth to understand whether any of this information is related to ASD development. This data will be updated monthly until each enrolled infant reaches 3 years of age, yielding a valuable compilation of information that will provide insight on how environmental changes affect whether the child develops ASD or not.

Microbiome: The human gut, compromised of the small and large intestine, is home to many types of bacteria. These bacteria help to break down and digest food, provide the body with energy, and make vitamins that the body need to thrive. This diverse community of bacteria is called the gut microbiome, which is known to play a large role in the development of the immune system. A main goal of the GEMMA study is to understand how the microbiome is affected by factors such as food intake or antibiotic drugs, and how this may affect the development of ASD. Investigators hope to learn more about this relationship by studying the members of the gut microbiome before and after autism development in the subset of enrolled infants who will develop ASD. The project will compare microbiota of ASD children with and without GI symptoms to determine whether different microbiota composition and differentially expressed bacterial genome perturb intestinal barrier function and immune response, leading to ASD in genetically at-risk infants. By doing this, the project will uncover patterns in the gut microbiome that may help investigators to predict who will develop ASD before it happens.

Metabolome: The processes that occur in the gut, such as the digestion of foods and production of vitamins, create products that are called metabolites. The specific metabolites that humans produce differ from person to person and depend on many factors, including genes, members of the gut microbiome, and food choices. The collection of metabolites produced by a sample is called the metabolome. The project will study the metabolomes of different infants while taking note of any changes to their environment and monitoring them for ASD. Studying the metabolites in this way is called metabolomics. In doing this, investigators hope to find patterns, or specific metabolomic profiles, that might predict when someone may develop ASD before it happens.

ELIGIBILITY:
Inclusion Criteria:

* Healthy newborns and infants less than 6 months of age who have not been introduced to solid foods (elementary formula feeding is permitted)
* First-degree relatives of ASD individuals (at least one sibling affected by ASD)

Exclusion Criteria:

* Infants older than 6 months of age
* Inability or unwillingness of legal guardian/representative to give written informed consent

Max Age: 6 Months | Sex: All
Age Groups: Child
Study Population: Newborns and infants less than 6 months of age who are first-degree relatives of ASD individuals (at least one sibling with an ASD diagnosis) are eligible for participation.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Use of microbiome/metagenomics/metatrancriptomic analysis to identify through our proposed prospective study and validate through large existing microbiome projects multi-omic biomarker predictors of ASD in at-risk infants. | 5 years
  i.e. stool and urine metabolites, alteration of gut permeability (via serum zonulin levels), abnormal immune response to dietary proteins (via IgA and IgG levels) and increased low-grade chronic inflammation (via serum pro-inflammatory cytokines).

CONTACTS AND LOCATIONS:
Overall Officials: Alessio Fasano, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- Massachusetts General Hospital for Children, Boston, Massachusetts, United States
- National University of Ireland Galway, Galway, Ireland
- The Azienda Sanitaria Locale Salerno, Salerno, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: GEMMA Study Website — https://www.gemma-project.eu/